CLINICAL TRIAL: NCT02667743
Title: Paclitaxel Micelles for Injection / Paclitaxel Injection in Combination With Cisplatin for First-line Therapy of Advanced NSCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Yizhong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM-03-2015
Record Dates: First submitted 2016-01-20; First posted 2016-01-29 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2020-03

CONDITIONS: Non-Small Cell Lung Cancer(NSCLC)
Keywords: NSCLC; Paclitaxel Micelles for Injection
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Injections; Paclitaxel; Cisplatin

ARMS (2):
- Paclitaxel Micelles for Injection + Cisplatin (Experimental): In the First Period, 230 mg/m2 of Paclitaxel Micelles for Injection was intravenously administrated for three hours without special infusion device, then 70 mg/m2 of Cisplatin was intravenously administrated for two hours. Three weeks constituted one course of treatment.
  In the Second Period, 300 mg/㎡ of Paclitaxel Micelles for Injection was intravenously administrated for three hours without special infusion device to patients whose minimum neutrophil ≥1.0 × 109 /L and minimum platelet count ≥80 × 109 /L and with no hematologic toxicity of grade II to IV occurred in the First Period. Then 70 mg/m2 of Cisplatin was intravenously administrated for two hours. Three weeks constituted one course of treatment.
  Interventions: Drug: Paclitaxel Micelles for Injection; Drug: Cisplatin
- Paclitaxel Injection + Cisplatin (Active Comparator): 175 mg/m2 of conventional Paclitaxel Injection was intravenously administrated for three hours, then 70 mg/m2 of Cisplatin was intravenously administrated for two hours. Three weeks constituted one course of treatment.
  Interventions: Drug: Paclitaxel Injection; Drug: Cisplatin

INTERVENTIONS:
Drug: Paclitaxel Micelles for Injection
  Arms: Paclitaxel Micelles for Injection + Cisplatin
Drug: Paclitaxel Injection
  Arms: Paclitaxel Injection + Cisplatin
Drug: Cisplatin

SUMMARY:
An open-label randomized and controlled clinical trial: This study was to compare the anticancer efficacy and safety in the First-Line Treatment in patients with Advanced Non-Small-Cell Lung Cancer with Paclitaxel Micelles for Injection In combination with Cisplatin versus Paclitaxel Injection Containing Cremophor EL(polyoxyethylenated castor oil) In combination with Cisplatin in the way of an open-label, randomized controlled clinical trial.

Treatment Protocol:

The subjects were randomized in the Paclitaxel Micelles for Injection Group and the Paclitaxel Injection Group by the proportion of 2:1. The centralized randomization method was adopted in this trial. Since the study was a comparison of first-line treatment, the test for superiority was adopted. The objective response rate was the primary indicator of efficacy in this study.

Trial Group:

Paclitaxel Micelles for Injection and Cisplatin was intravenously administrated. Three weeks constituted one course of treatment.

No pretreatment, including anti-allergic prevention and antiemetic prophylaxis, was required for the patients before infusion of Paclitaxel Micelles for Injection patients.

Control Group:

Conventional Paclitaxel Injection and Cisplatin was intravenously administrated. Three weeks constituted one course of treatment.

Standard preventive treatment must be given to patients in accordance with the specific requirements in specifications of Paclitaxel Injection.

Regardless of the Trial Group or the Control Group, six treatment periods shall be the upper limit.

To estimate the sample size based on objective remission indicators (CR + PR) in the study. Hypothesis: the objective remission rate of the Paclitaxel Micelles for Injection combined with Cisplatin in the Trial Group is different with that of first-line treatment of advanced non-small cell lung cancer, and is also different with that of the Cremophor EL-containing Paclitaxel Injection combined with Cisplatin in the Control Group. Trial parameter settings: assuming α = 0.05 and 1-β = 80%, the Trial Group: Control Group is designed as per the proportion of 2: 1. According to the sample size formula , a total of 426 patients is required, including 284 patients assigned in the Trial Group and 142 in the Control Group. In consideration of case expulsion in the process of clinical, enlarged by 10%, actually 468 cases were included in the groups, including 312 in the Trial Group and 156 in the Control Group.

ELIGIBILITY:
Inclusion Criteria:

1. First-line patients with locally advanced or metastatic NSCLC (Clinical Stage of ⅢB/Ⅳ, TNM (primary tumor, regional nodes, metastasis) Staging Edition 7) confirmed by histological or cytological diagnosis or of postoperative recurrence;

   First-line patients include:
   1. Patients who are newly diagnosed as ⅢB/Ⅳ and have undergone no radiotherapy or chemotherapy or molecular targeting treatment;
   2. Patients with postoperative reoccurrence and metastasis and receiving no adjuvant radiotherapy or chemotherapy or molecular targeting treatment;
   3. Patients with postoperative reoccurrence and metastasis and receiving adjuvant radiotherapy or chemotherapy or molecular targeting treatment, but it has been more than one year since the end of such therapies or treatment.
   4. Patients who have received prior radiotherapy can be enrolled. However, the radiation area must be <25% of bone marrow area, the prior radiotherapy has been completed at least 4 weeks before the enrollment, and the acute radiation toxicity must have been restored. Local lesions that have undergone radiotherapy are not allowed to be included in the measurable lesions save as such lesions with significant progress recorded after the last radiotherapy.
2. Patients with available measurable lesions in line with the requirements of "measurable lesions" in the response evaluation criteria "RECIST Version 1.1". Lesions with at least one accurately measurable diameter (serve as the maximum diameter): the maximum diameter of target lesions with CT scan ≥20 mm or the maximum diameter with spiral CT or MRI scan ≥10 mm;
3. ECOG (Eastern Cooperative Oncology Group) score ≤ 1 points and expected survival of at least 3 months;
4. 18 to 70 years old, male or female;
5. Blood picture and functions of major organs such as heart, lung, liver, kidneys are basically normal.
6. Blood routine test must meet the following criteria:

   1. ANC≥1.5×109/L；
   2. PLT≥100×109/L；
   3. Hb≥90g/L。
7. Blood biochemical test must meet the following criteria:

   1. Plasma total bilirubin ≤1.5 × upper limit of normal (ULN);
   2. ALT (Alanine aminotransferase), AST (Aspartate transaminase) or AKP≤2.5 × ULN (for patients with hepatic metastases, ALT, AST or AKP≤5 × ULN; for patients with bone metastases, AKP≤10 × ULN);
   3. Cr ≤1.5 × ULN;
8. Patients have no cardiac insufficiency symptoms at baseline; no serious abnormal signs in ECG
9. Efficacy of cancer-related imaging examinations are completed within 2 weeks before enrollment and clinical condition assessment, the three routine tests of blood, urea, and stool, blood biochemical examination, ECG, CEA (carcinoembryonic antigen) and other examinations completed within 1 week before enrollment;
10. Patients can understand the purpose of the clinical trial, participate out of their own will, and sign the informed consent;
11. Patients have good compliance, accept the doctor's follow-up evaluations, and voluntarily follow treatment protocol during the study;
12. Male or female patients with childbearing potential voluntarily take contraceptive measures during the trial.

Exclusion Criteria:

In case of any of the following circumstances, the patient is not allowed to participate in this study:

1. Patients known to have mutant EGFR (epidermal growth factor receptor), ALK (anaplastic lymphoma kinase) in genetic examinations;
2. Patients with primary brain or central nervous metastases (including leptomeningeal metastasis), excluding patients with asymptomatic single brain metastasis under strict control; and patients with central nervous tumors accompanied by cerebral hypertension or neuropsychiatric symptoms;
3. Patients with non-eliminated acute and chronic infections or patients also suffer from other serious diseases simultaneously;
4. Patients who cannot complete the entire trial process as the investigator may deem fit;
5. Patients with peripheral neuropathy above grade I;
6. Patients with an allergic history to Paclitaxel;
7. The existence of a third space effusion that cannot be controlled by drainage or other means (such as middle - large pleural effusion, middle - large pericardial effusion and ascites); patients with asymptomatic small pleural effusion requiring no clinical intervention may be enrolled subject to strict control;
8. Patients with mental illness or mental disorders, poor compliance, or cannot account treatment responses;
9. Patients with poor tolerability due to serious organic diseases or major organ failure, such as decompensated heart and lung failure;
10. Patients with bleeding tendency diseases;
11. Organ transplant recipients;
12. Patients with drug abuse and other adverse drug addicts, long-term alcoholics and patients with AIDS and other infectious diseases;
13. Long-term users of adrenal corticosteroids or immunosuppressive agents;
14. Patients have suffered from other malignant cancers within 5 years (except for cured basal cell carcinoma and cervical carcinoma in situ);
15. Patients with active hepatitis and liver metastasis exceeding three-quarters of the whole liver.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Baseline to measured PD (up to 36 months)
  Objective response rate is defined as the proportion of subjects with complete or partial response as determined by the investigator using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)

SECONDARY OUTCOMES:
Progression-Free-Survival | Randomization to measured PD or date of death from any cause (up to 36 months)
  PFS(Progression-Free-Survival) was the time from randomization until the date of objectively determined progressive disease (PD) or death due to any cause, whichever occurred first.
Overall survival | Randomization to date of death from any cause (up to 36 months)
  Overall survival was the time from randomization until the date of death from any cause. Participants who were alive at the end of the follow-up period (or lost to follow-up) were censored on the last date the participant was known to be alive.
Incidence of Adverse Events，Serious Adverse Events. | up to 36 months
Incidence of bone marrow suppression. | up to 36 months
The number of patients with dose adjustment. | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, Principal Investigator — Shanghai Chest Hospital; Yilong Wu, Principal Investigator — Guangdong Provincial People's Hospital; Meiqi Shi, Principal Investigator — Jiangsu Cancer Institute & Hospital
Locations (3):
- China (3):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Jiangsu Cancer Hospital, Nanjing, Zhejiang

REFERENCES:
- [Derived] Shi M, Gu A, Tu H, Huang C, Wang H, Yu Z, Wang X, Cao L, Shu Y, Wang H, Yang R, Li X, Chang J, Hu Y, Shen P, Hu Y, Guo Z, Tao M, Zhang Y, Liu X, Sun Q, Zhang X, Jiang Z, Zhao J, Chen F, Yu H, Zhang W, Sun J, Li D, Zhou J, Han B, Wu YL. Comparing nanoparticle polymeric micellar paclitaxel and solvent-based paclitaxel as first-line treatment of advanced non-small-cell lung cancer: an open-label, randomized, multicenter, phase III trial. Ann Oncol. 2021 Jan;32(1):85-96. doi: 10.1016/j.annonc.2020.10.479. Epub 2020 Oct 29. PMID 33130217